CLINICAL TRIAL: NCT00425958
Title: Examination of Virtual Supermarket (Vmall) as an Assessment of Executive Functions in Children and Adolescents With Acquired Brain Injury
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA-05-3856-AB-CTIL
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2007-09-26 (Estimated); Status verified 2007-09

CONDITIONS: Brain Injuries
Keywords: year and more after TBI; good vision; at least one functinal hand; cap[able od doing shopping during everyday life
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research is to find whether or not there are differences in the executive functions during "shopping" in a "virtual mall", between children with Acquired Brain Injury (ABI) vs healthy children.

The hypothesis is that there will be differences in time (more time to shop) and mistakes (more mistakes during shopping), in the ABI group.

ELIGIBILITY:
Inclusion Criteria:

* children with ABI
* at least a year after injury
* who have been discharged from hospital and back home

Exclusion Criteria:

* children with learning disabilities former to injury
* visual disabilities or developmental disabilities

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2006-04; Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amichai Brezner, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel